CLINICAL TRIAL: NCT04202367
Title: Transversus Abdominis Plane (TAP) Block With Different Bupivacaine Concentrations in Pediatric Patients Undergoing Unilateral Inguinal Hernia Repair Surgery: A Prospective Randomised Double-Blinded Study
Brief Title: The Efficacy of Different Bupivacaine Concentrations in Pediatric Patients Undergoing Transversus Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/1281
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Transversus Abdominis Plane Block
Keywords: Transversus abdominis plane block; Bupivacaine; Concentration; Postoperative analgesia; Inguinal hernia repair surgery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Ultrasound-guided TAP block was applied following standard general anaesthesia induction. All patients received remifentanil 0,1 μg/kg/h infusion and paracetamol 15 mg/kg intraoperatively, and paracetamol 4x15 mg/kg per day postoperatively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Seventy-four patients aging between 1 and 8 years, undergoing unilateral inguinal hernia surgery, were enrolled in the study and were randomized using closed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block with 1 mg.kg-1 bupivacaine 0.25% (Active Comparator): Patients had 1 mg.kg-1 bupivacaine 0.25% with US-guided TAP block
  Interventions: Drug: 1 mg.kg-1 bupivacaine 0.25%
- TAP block with 1 mg.kg-1 bupivacaine 0.125% (Active Comparator): Patients had 1 mg.kg-1 bupivacaine 0.125% with US-guided TAP block
  Interventions: Drug: 1 mg.kg-1 bupivacaine 0.125%

INTERVENTIONS:
Drug: 1 mg.kg-1 bupivacaine 0.25% — Ultrasound-guided transversus abdominis plane block for unilateral inguinal hernia repair surgery.
  Other Names: Marcaine
  Arms: TAP block with 1 mg.kg-1 bupivacaine 0.25%
Drug: 1 mg.kg-1 bupivacaine 0.125% — Ultrasound-guided transversus abdominis plane block for unilateral inguinal hernia repair surgery.
  Other Names: Marcaine
  Arms: TAP block with 1 mg.kg-1 bupivacaine 0.125%

SUMMARY:
This study is designed to compare the analgesic efficacy of different bupivacaine concentrations in pediatric patients undergoing ultrasound-guided transversus abdominis plane (TAP) block for unilateral inguinal hernia repair. In recruited 74 patients; Group 1 (n:37) received 1 mg/kg bupivakain 0.25% and Group 2 (n: 37) received 1 mg/kg bupivakain 0.125% for ultrasound-guided TAP block following standard general anaesthesia induction. FLACC (Face, Legs, Activity, Cry, Consolability) behavioral pain assessment scale was used for evaluating patients' postoperative pain levels at 15-, 30-, 45-minute and 1-, 2-, 6-, 24-hour. Tramadol 1 mg/kg was administered intravenously as rescue analgesic when FLACC score was ≥4. Total analgesic requirement, length of hospital stay and side effects were recorded.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block is a safe and effective analgesia technique for paediatric patients. This study is designed to compare the analgesic efficacy of different bupivacaine concentrations in paediatric patients undergoing ultrasound-guided TAP blocks for unilateral inguinal hernia repair surgery. Seventy-four patients aging between 1 and 8 years, undergoing unilateral inguinal hernia surgery, were enrolled for this study after obtaining Institutional Ethics Committee approval and written informed consents from parents or legal guardians (2016/1281). Group 1 (n:37) received 1 mg/kg bupivakain 0.25% and Group 2 (n: 37) received 1 mg/kg bupivakain 0.125% for ultrasound-guided TAP block following standard general anaesthesia induction. All patients received remifentanil 0,1 μg/kg/h infusion and paracetamol 15 mg/kg intraoperatively, and paracetamol 4x15 mg/kg per day postoperatively. FLACC (Face, Legs, Activity, Cry, Consolability) behavioral pain assessment scale was used for evaluating patients' postoperative pain levels at 15-, 30-, 45-minute and 1-, 2-, 6-, 24-hour. Tramadol 1 mg/kg was administered intravenously as rescue analgesic when FLACC score was ≥4. Total analgesic requirement, length of hospital stay and side effects were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status I/II
* Children between 1 to 8 years of age
* Patients undergoing unilateral inguinal hernia repair surgery

Exclusion Criteria:

* Denial of parents
* Patients who are allergic to local anesthetics

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
FLACC pediatric pain scores | up to 24 hours
  It corporates five categories of behavior, each scored on 0-2 point scale so that total score ranges from 0-10.

SECONDARY OUTCOMES:
Total analgesic requirement | up to 24 hours
  Tramadol
First analgesic requirement time | up to 24 hours
  Duration of postoperative analgesia
Incidence of side effects | up to 24 hours
  Nausea, vomiting, respiratory depression
The length of hospital stay | up to 24 hours
  Hospitalisation hours
Incidence of complications | up to first week.
  Hemotoma, infection

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Assoc. Prof, Principal Investigator — Istanbul University; Emine Aysu Salviz, Assoc. Prof, Study Chair — Istanbul University

REFERENCES:
- [Derived] Karadeniz MS, Atasever AG, Salviz EA, Bingul ES, Ciftci HS, Dincer MB, Sungur MO. Transversus abdominis plane block with different bupivacaine concentrations in children undergoing unilateral inguinal hernia repair: a single-blind randomized clinical trial. BMC Anesthesiol. 2022 Nov 21;22(1):355. doi: 10.1186/s12871-022-01907-y. PMID 36411426